CLINICAL TRIAL: NCT02281565
Title: Knowledge, Attitude and Practice About Blood Donation Among Medical Students and Medical Staff
Brief Title: Attitudes About Blood Donation
Acronym: KAPsurvey
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: International Institute of Rescue Research and Education (Other)
Responsible Party: Principal Investigator, Lukasz Szarpak, Lukasz Szarpak, International Institute of Rescue Research and Education
Other Study IDs: Blood_donation2014
Record Dates: First submitted 2014-10-27; First posted 2014-11-03 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Blood Donation
Keywords: attitudes; blood donation; blood shortage
MeSH Terms: conditions — Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: survey — Survey about Knowledge, Attitude and Practice About Blood Donation

SUMMARY:
The study evaluates the knowledge, attitude and practice about blood donation among medical students and medical staff in Poland.

DETAILED DESCRIPTION:
In Poland, the blood gives an average of 31 people per 1.000 inhabitants, while in Western Europe the rate was twice as high.

In the study the investigators are examining how medical students and medical staff feel about the issues of blood donation, especially: blood shortage.

The investigators are planning to focus on the following specific questions:

What is the level of knowledge about blood donation among participants? What are the sociodemographic, sociocultural and socioeconomic characteristics of blood donors and non-blood donors among medical staff and medical students? Evidence on the role of financial and other incentives in eliciting blood donation.

ELIGIBILITY:
Inclusion Criteria:

* Give voluntary consent to participate in the study

Exclusion Criteria:

* not meet the above criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Medical staff: medical doctors, nurses, paramedics Medical students: PhD students, medicine students, nursing and paramedics studies
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-10; Primary Completion 2014-11 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who approve prosocial motivation to blood donation | 3 months
  Percentage of healthcare workers and medical students with appropriate attitude assessed by 10- items questionnaire about perception towards financial and other incentives in eliciting blood donation. For each correct answer participant receive 1 point (0-1 point scale).

SECONDARY OUTCOMES:
Results of the Medical Knowledge Tool (Questionnaire) | 3 months
  Percentage of healthcare workers and medical students with appropriate knowledge assessed by 10- items questionnaire about basic information about blood donation standards and registry. For each correct answer participant receive 1 point (0-1 point scale).
Results of the Practice Tool (Questionnaire) | 3 months
  Percentage of healthcare workers and medical students with appropriate practice assessed by 10- items questionnaire about basic information about practice with blood donation (prohibited and unethical practices). For each correct answer participant receive 1 point (0-1 point scale).

CONTACTS AND LOCATIONS:
Locations (1):
- International Institute of Rescue Research and Education, Warsaw, Masovia, Poland